CLINICAL TRIAL: NCT03863730
Title: Profermin®: Prevention of Progression in Alcoholic Liver Disease by Modulating Dysbiotic Microbiota - a Randomized Controlled Clinical Trial
Brief Title: Profermin®: Prevention of Progression in Alcoholic Liver Disease by Modulating Dysbiotic Microbiota
Acronym: SYN-ALD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); University of Southern Denmark (Other); Nordisk Rebalance A/S (Industry)
Responsible Party: Principal Investigator, Aleksander Krag, Professor, PhD, Cand.Med., Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20170163
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Alcoholic Liver Disease; Liver Cirrhosis, Alcoholic; Probiotics; Liver Fibrosis
Keywords: Food for special medical purposes; Gut and liver axis
MeSH Terms: conditions — Liver Diseases, Alcoholic; Liver Cirrhosis, Alcoholic; Liver Cirrhosis | interventions — Probiotics; Fresubin; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive Profermin Plus® versus a general FSMP, Fresubin®, for 24 weeks.
Masking Description: Pathologist will perform outcome assessment blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Profermin Plus® (Experimental): Intervention group will be drinking the liver-specialized product Profermin Plus®, based on fermented oats, Lactobacillus Plantarum 299v, barley malt and lecithin. The product also contains Thiamin, which is beneficial in patients with liver diseases.
  Interventions: Dietary Supplement: Profermin Plus, FSMP, probiotics
- Fresubin® (Active Comparator): Fresubin® is a standard FSMP and will be used as control product. Since Profermin Plus® is a disease-specific FSMP, the documentation must prove an effect that cannot be achieved by modification of the normal diet alone or by standard FSMP's. Therefor the comparator must be a standard FSMP, i.e. a nutritionally complete FSMP with standard nutrient formulation, which may constitute the sole source of nourishment of a person, hence the reason for using Fresubin® as comparator.
  Interventions: Dietary Supplement: Fresubin, dietary supplement

INTERVENTIONS:
Dietary Supplement: Profermin Plus, FSMP, probiotics — Participants will have to supply their normal intake with Profermin Plus, FSMP, Prbiotics product twice every day for 24 weeks.
  The product Profermin Plus® has changed its name to ReFerm®. The content of the product is unchanged. The change occurred after the clinical part of the study was completed.
  Arms: Profermin Plus®
Dietary Supplement: Fresubin, dietary supplement — Participants will have to supply their normal intake with the control product, Fresubin, dietary supplement twice every day for 24 weeks.
  Arms: Fresubin®

SUMMARY:
Investigators wishes to influence the gut microbiota in patients with alcoholic liver disease in a randomized controlled clinical trial. The investigators hypothesize that the alcohol-related dysbiosis seen in these patients can be changed and disease progression haltered by modulating microbiota with probiotics during 24 weeks.

DETAILED DESCRIPTION:
Chronic alcohol overuse is associated with increased gut permeability and in addition, the intestinal microbiota changes qualitatively (dysbiosis) and quantitatively (bacterial overgrowth) in alcoholic liver disease in favour of a microbiota with increased invasive potential. As a consequence, an increased load of bacterial products is transported to the liver leading to inflammation and fibrogenesis.

This cross talk between the intestinal microbiota and the liver constitute a gut-liver axis, which is increasingly recognized as key mechanism in the progression of liver disease and pathogenesis of liver related complications.

The investigators hypothesize that the gut microbiota and its metabolites are major drivers of fibrosis in human liver disease and that modulating the intestinal flora by Profermin® (a food for special medical purposes) will modulate the alcohol related dysbiotic signatures in the microbiota which may halter disease progression by reducing activity of hepatic stellate cells.

Dietary supplements that alter the microbiome towards a more beneficent type may improve liver inflammation and thus be a better alternative than supplements that simply add nutrients. Investigators expect that the trial will provide proof-of-concept for a sustainable dietary strategy in liver fibrosis.

Examples of biopsies which did not meet quality criteria for reliable histological reading, led to inclusion of 16 extra patients. In total we included 56 patients to ensure an adequate number of participants with valid liver biopsy data for assessment of the primary endpoint and intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Prior or ongoing harmful alcohol intake defined as an average of ≥24g alcohol/day for women and ≥36g/d for men for ≥ 5 year.

  * Outpatients with compensated advanced chronic alcohol-related liver disease, defined as stable patients with:

    1. liver stiffness ≥15 kPa and asymptomatic and/or
    2. New liver biopsy (<6months) with at least F3 fibrosis (kleiner) and/or
    3. Liver biopsy older that 6 months with liver stiffness ≥10 kPa
  * Understand and speak Danish written and orally
  * Informed consent

Exclusion Criteria:

* Hospitalised
* Moderete or severe Ascites, determined from imaging diagnostics
* High-risk varices needing interventional treatment (endoscopy, TIPS)
* Child-Pugh C score
* MELD-Na ≥15
* Lactose intolerance
* Coeliac disease
* Irritable bowel syndrome defined by ROME III criteria
* Antibiotic treatment the prior 3 months
* Treatment with nutritional drinks, probiotics or prebiotics within the last 3 months
* The investigator judge that the patient would not be compliant with trial medicine
* Pregnancy
* Known liver disease other than alcoholic, of any aetiology
* Severe malnutrition
* Malignancy - except spino- or basocellular skin cancer. Patients with prior malignant disease are allowed if cancer-free for at least one year
* Recent infectious gastroenteritis (for the last 6 weeks)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Hepatic stellate cell activity | 24 weeks
  Attenuation of liver hepatic stellate cell activity, defined as the proportion of patients with a 10% or more reduction in activated hepatic stellate cells, measured by a-smooth muscle actin (a-SMA) stain quantification of liver biopsies.

SECONDARY OUTCOMES:
Hepatic a-SMA activity | 24 weeks
  Reduction in hepatic a-SMA activity
Hepatic inflammation | 24 weeks
  Evaluated by hepatic inflammation markers and metabolites
Alfa-smooth muscle actin concentration | 24 weeks
  Reduction in circulating a-smooth muscle actin concentration
Hepatic venous pressure gradient (HVPG) | 24 weeks
  Reduction in portal pressure measured by the HVPG in unit mmhg
Reduction in non-invasive fibrosis markers | 24 weeks
  Reduction in Ultrasound shear wave elastography (transient and 2-dimensional) (kPa)
Reduction in non-invasive fibrosis markers | 24 weeks
  ProC3 and ProC4 (ng/ml)
Reduction in non-invasive fibrosis markers | 24 weeks
  ELF test
Reduction in non-invasive fibrosis markers | 24 weeks
  Forns index
Reduction in non-invasive fibrosis marker | 24 weeks
  APRI score
Reduction in non-invasive fibrosis markers | 24 weeks
  FIB4 (points)
Markers of liver inflammation | 24 weeks
  Reduction in circulating markers of liver inflammation (cytokeratin-18 degradation products M30 and M65)
Improvement of liver histological lesions | 24 weeks
  Improvement in semiquantitative liver histological lesions that fulfil at least one of two criteria:
  * At least one stage of liver fibrosis improvement according to the Kleiner fibroses classification (0-4), with no worsening of hepatic inflammatory activity
  * Complete resolution of hepatic inflammatory activity, with no worsening of fibrosis.
  [Worsening defined as an increase of at least one stage of either lobular inflammation or hepatocyte ballooning. Resolution defined as ballooning=0 and lobular inflammation=0-1]
Improvement in gut dysbiosis | 24 weeks
  Defined as:
  * Improved taxonomy, defined as increased relative abundance of species characteristic of healthy individuals and decreased relative abundance of species characteristic of cirrhosis and severe alcoholic liver disease
  * Increase in gut microbial richness
Liver vein outflow of microbial products | 24 weeks
  Change in Liver vein outflow of microbial products
Lipid profile | 24 weeks
  Improvement of lipid profile defined as:
  Rising HDL, decrease in triglycerids, LDL and total cholesterol
Any changes in non-invasive markers of steatosis | 24 weeks
  Controlled Attenuation Parameter(CAP) and ultrasonographic steatosis assessment (bright liver echo pattern)
Individual domains of NAS scoring systemt | 24 weeks
  Any changes in individual domains of the NAS scoring system (fibrosis 0-4, steatosis 0-3, lobular inflammation 0-2, portal inflammation 0-1, ballooning 0-2) or in collagen proportionate area (%)
Metabolic changes | 24 weeks
  Water soluble metabolites in circulation will be evaluated with metabolomics
Changes in circulating cytokines | 24 weeks
  Cytokines related to cardiovascular disease and inflammation will be analysed
Changes in hepatic macrophage activity | 24 weeks
  Changes in digital imaging analysis of hepatic CD163 expression in liver biopsies
Changes in intestinal fibrosis markers | 24 weeks
  C4M generated by decomposition of type 4 collagen
Changes in intestinal fibrosis markers | 24 weeks
  CPA9-HNE a fragment degraded from calprotectin
Changes bile acids | 24 weeks
  Changes in bile acids will be measured in both stool and circulation
Metabolic changes | 24 weeks
  Amino acids in circulation will be evaluated with metabolomics
Metabolic changes | 24 weeks
  Lipidomics in circulation will be evaluated with metabolomics
Metabolic changes | 24 weeks
  Lipidomics in liver samples will be evaluated with metabolomics
Metabolic changes | 24 weeks
  Short chain fatty acids in circulation will be evaluated with metabolomics
Metabolic changes | 24 weeks
  Short chain fatty acids in stool samples will be evaluated with metabolomics

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - FLASH - Centre of Liver Research, Odense, Fyn
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No